CLINICAL TRIAL: NCT00061139
Title: Randomized Controlled Trial of Pediatric CI Therapy
Brief Title: Constraint-Based Therapy to Improve Motor Function in Children With Cerebral Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD040692 (NIH)
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Cerebral Palsy; Motor Deficits
Keywords: Cerebral palsy; Hemiparesis; Pediatric CI therapy; Upper extremity; Training; Limb restraint
MeSH Terms: conditions — Cerebral Palsy; Neurologic Manifestations; Paresis

INTERVENTIONS:
Behavioral: Pediatric Constraint-Induced Movement therapy
Behavioral: Conventional pediatric motor rehabilitation therapy

SUMMARY:
Pediatric Constraint-Induced (CI) Movement therapy is a rehabilitation program designed to improve motor function in children with partial paralysis. Children with cerebral palsy may have one arm that has significantly greater function (good arm) than the other (bad arm). Restricting the use of the good arm may improve the use of the bad arm. In pediatric CI therapy, the good arm is put in a sling to force increased use of the bad arm. The bad arm is also trained each day for several weeks. This study will test the ability of pediatric CI therapy to improve motor function in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy afflicts at least two in 1,000 children in the United States and approximately 2,000,000 children worldwide. Behavioral techniques that impact the plasticity of the nervous system need to be incorporated into practical, evidence-based therapeutic interventions for this condition.

CI therapy was derived from basic research with animal and human subjects. Randomized, controlled studies indicate that it can substantially reduce the motor deficit of adult patients with mild to moderately severe chronic strokes and can increase their independence over a period of years. CI therapy involves motor restriction of the less affected upper extremity for a period of 2 to 3 weeks while concurrently training the more affected upper limb. This gives rise to concentrated, repetitive use of the more affected extremity. In adults, CI therapy has lead to a large increase in use-dependent cortical reorganization involving the recruitment of substantial new regions of the brain in the innervation of more affected extremity movement.

The study will evaluate CI therapy in a pediatric population. The study will test whether pediatric CI therapy can promote new and improved motor behavior in young children with hemiparesis associated with cerebral palsy. Pediatric CI therapy involves total restraint of the unaffected upper extremity with simultaneous repetitive use of the affected extremity for 6 hours/day for 21 consecutive days.

Fifty-two children ages 2 to 6 years old with hemiparetic cerebral palsy will be randomly assigned to either the pediatric CI therapy group or to a control group. The control group will receive standard rehabilitation therapy. All children will have a complete medical evaluation with emphasis on motor function prior to treatment initiation. Children will undergo follow-up testing at 1, 6, and 12 months post-treatment. The primary study assessment tools are the Pediatric Developmental Motor Scales - II (PDMS-II), DASI - II, Bayley Developmental Skills Test, Pediatric Motor Activity Log (PMAL), Child Arm Use Test (CAUT), and Emerging Behavior Scale (EBS).

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of hemiparetic cerebral palsy consistent with criteria in Swaiman and Russman (1999) and Badawi et al. (1998)
* Recommended for participation in pediatric rehabilitation and/or early intervention
* Lives within 50 miles of the Civitan Center at University of Alabama at Birmingham or the family is willing to temporarily relocate to the Birmingham area for treatment

Exclusion Criteria

* Profound bilateral hearing loss with the use of hearing aids
* Severe visual impairment
* Serious seizure disorder or uncontrolled seizures
* Genetic and syndromic conditions historically excluded for CP registries
* Familial Spastic Paraplegia
* Ataxic Cerebral Palsy
* Diagnosis of Pervasive Developmental Disability or autism
* Serious or recurring medical complications
* Scheduled for surgery within 12 months of study entry

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52
Dates: Start 2002-09; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Edward Taub, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States